CLINICAL TRIAL: NCT05263908
Title: General Investigation for PAXLOVID PAC
Brief Title: A Study to Learn About PAXLOVID (a Commercial Medicine) In People With COVID-19
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4671018; NCT05263908 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-02-25; First posted 2022-03-03 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: SARS-CoV-2 Infection
Keywords: severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); coronavirus disease 2019 (COVID-19); Paxlovid; Nirmatrelvir
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PAXLOVID PACK: Subjects administered PAXLOVID PACK
  Interventions: Drug: nirmatrelvir / ritonavir

INTERVENTIONS:
Drug: nirmatrelvir / ritonavir — The usual dosage in adults and pediatric patients (≥12 years of age weighing ≥40 kg) is 300 mg of Nirmatrelvir and 100 mg of ritonavir all taken together orally twice daily for 5 days.
  Other Names: PAXLOVID PACK

SUMMARY:
The purpose of this post marketing observational study is to learn about the safety and effects of the commercial medicine (called PAXLOVID) for the treatment of COVID-19. This study is intended to be registered with the participants who:

* Have taken PAXLOVID PACK and have no history of using this medicine.
* Are 12 years and older

All participants will receive PAXLOVID, a standard treatment for COVID-19. Participants will take PAXLOVID 2 times a day by mouth or as prescribed.

We will examine the experiences of people taking PAXLOVID. This will help us determine if PAXLOVID is safe and effective.

Participants will be followed up for 28 days after taking PAXLOVID. During this time, participants will be closely watched for the safety and effects of PAXLOVID.

DETAILED DESCRIPTION:
This is a multicenter cohort study to be conducted in individuals with SARS-CoV-2 infection who are treated with this product, and the investigator will enter the information required in this study in the case report forms (CRFs) based on the information obtained through medical records.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are administered PAXLOVID PACK and have no history of using this drug.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects who have been treated with PAXLOVID PACK for the first time.
Sampling Method: Probability Sample
Enrollment: 3346 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local County, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Murata K, Hyokai S, Fujii Y, Morimasa M. Real-world safety of nirmatrelvir plus ritonavir in patients with COVID-19 in Japan: A post-marketing surveillance study. Jpn J Infect Dis. 2026 Jan 30. doi: 10.7883/yoken.JJID.2024.380. Online ahead of print. PMID 41621946
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671018

RESULTS

PARTICIPANT FLOW:
Groups:
- Paxlovid PACK (Nirmatrelvir/Ritonavir): Participants who received Paxlovid PACK as indicated in the approved local product document for the first time were observed from the start date of treatment with Paxlovid PACK to 28 days after the end of treatment (the day following the end of treatment was defined as Day 1). The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Paxlovid PACK (Nirmatrelvir/Ritonavir)
Started | 3346
Completed | 2948
Not Completed | 398
Not completed — No informed consent for publication of study results | 397
Not completed — CRF not collected | 1

BASELINE CHARACTERISTICS:
Population: A total of 2948 participants completed the study. Of the 2948 participants, 119 participants were excluded from the safety analysis set due to the following reasons: no information on administration (13 participants), no information on adverse events - no re-visits (106 participants). Overall, the safety analysis set comprised of 2829 participants.
Arm/Group | Paxlovid PACK (Nirmatrelvir/Ritonavir)
Number analyzed (Participants) | 2829
Age, Customized [Number; unit: Participants]
  <15 years | 2
  ≥15 and <65 years | 1404
  ≥65 years | 1423
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1324
  Male | 1505
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Drug Reactions
Description: Adverse drug reaction (ADR) was a treatment-related adverse event and any untoward medical occurrence attributed to Paxlovid PACK in a participant who received Paxlovid PACK. Serious adverse drug reaction (SADR) was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Relatedness to Paxlovid PACK was assessed by the physician.
Time Frame: From the start date of treatment with Paxlovid PACK to 28 days after the end of treatment, up to approximately 45 days.
Population: The safety analysis set (2829 participants) comprised of participants who satisfied the inclusion criteria. Participants with no informed consent for publication of study results, no information on administration, and no information on adverse events - no re-visits were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Paxlovid PACK (Nirmatrelvir/Ritonavir)
Number analyzed (Participants) | 2829
Participants
  ADR | 423
  SADR | 6

2. Secondary Outcome: Percentage of Participants With Worsening Severity (Efficacy Analysis Set #1)
Description: Whether the severity of infection caused by SARS-CoV-2 had worsened was evaluated.
  However, when the severity was severe at the start of Paxlovid PACK and did not worsen during the observation period, it was considered as "severe at the start of treatment."
Time Frame: From the start date of treatment with Paxlovid PACK to 28 days after the end of treatment, up to approximately 45 days.
Population: For the efficacy analysis set #1 (2828 participants), participant with disease not subject to the study (1 participant) was excluded from the safety analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paxlovid PACK (Nirmatrelvir/Ritonavir)
Number analyzed (Participants) | 2828
Percentage of participants
  Worsened | 2.19 [1.68 to 2.80]
  Not worsened | 94.77 [NA to NA] — The 95% Confidence Interval was not calculated.
  Severe at the start of treatment | 0 [NA to NA] — The 95% Confidence Interval was not calculated.
  Unknown (worsening unknown) | 3.04 [NA to NA] — The 95% Confidence Interval was not calculated.

3. Secondary Outcome: Percentage of Participants With Worsening Severity (Efficacy Analysis Set #2)
Description: as for outcome 2
Time Frame: From the start date of treatment with Paxlovid PACK to 28 days after the end of treatment, up to approximately 35 days.
Population: For the efficacy analysis set #2 (1965 participants), participants other than outpatient at the start of treatment (863 participants) were excluded from the efficacy analysis set #1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paxlovid PACK (Nirmatrelvir/Ritonavir)
Number analyzed (Participants) | 1965
Percentage of participants
  Worsened | 1.63 [1.12 to 2.29]
  Not worsened | 94.66 [NA to NA] — The 95% Confidence Interval was not calculated.
  Severe at the start of treatment | 0 [NA to NA] — The 95% Confidence Interval was not calculated.
  Unknown (worsening unknown) | 3.72 [NA to NA] — The 95% Confidence Interval was not calculated.

4. Secondary Outcome: Percentage of Participants With Worsening Severity (Efficacy Analysis Set #3)
Description: as for outcome 2
Time Frame: From the start date of treatment with Paxlovid PACK to 28 days after the end of treatment, up to approximately 35 days.
Population: For the efficacy analysis set #3 (1905 participants), participants with no risk factors of progressing to severe illness (60 participants) were excluded from the efficacy analysis set #2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paxlovid PACK (Nirmatrelvir/Ritonavir)
Number analyzed (Participants) | 1905
Percentage of participants
  Worsened | 1.68 [1.15 to 2.36]
  Not worsened | 94.59 [NA to NA] — The 95% Confidence Interval was not calculated.
  Severe at the start of treatment | 0 [NA to NA] — The 95% Confidence Interval was not calculated.
  Unknown (worsening unknown) | 3.73 [NA to NA] — The 95% Confidence Interval was not calculated.

5. Secondary Outcome: Cumulative Incidence Rate of COVID-19 Related Hospitalization or Death From Any Cause Through Day 28 (Efficacy Analysis Set #3)
Description: The percent probability is the percent of the participants who had COVID-19 related hospitalization or death from any cause.
Time Frame: 3, 5, 7, 14, 21 and 28 days after the start of administration with Paxlovid PACK.
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Paxlovid PACK (Nirmatrelvir/Ritonavir)
Number analyzed (Participants) | 1905
Percent probability
  3 days from the start of administration of this drug | 3.99 [3.20 to 4.97]
  5 days from the start of administration of this drug | 4.41 [3.58 to 5.44]
  7 days from the start of administration of this drug | 4.47 [3.63 to 5.50]
  14 days from the start of administration of this drug | 4.80 [3.93 to 5.87]
  21 days from the start of administration of this drug | 4.86 [3.98 to 5.93]
  28 days from the start of administration of this drug | 4.92 [4.03 to 6.00]

6. Secondary Outcome: Cumulative Incidence Rate of COVID-19 Related Hospitalization or Death From Any Cause Through Day 28 (Sensitivity Analysis) (Efficacy Analysis Set #3)
Description: The percent probability is the percent of the participants who had COVID-19 related hospitalization or death from any cause.
  Sensitivity analysis was conducted by changing the event definition of "hospitalization for treatment of infection caused by SARS-CoV-2" as follows: there were concomitant medications for infection caused by SARS-CoV-2 or concomitant non-drug therapies due to infection caused by SARS-CoV-2 on or after the date of administration.
Time Frame: 3, 5, 7, 14, 21 and 28 days after the start of administration with Paxlovid PACK.
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Paxlovid PACK (Nirmatrelvir/Ritonavir)
Number analyzed (Participants) | 1905
Percent probability
  3 days from the start of administration of this drug | 1.42 [0.97 to 2.06]
  5 days from the start of administration of this drug | 1.58 [1.11 to 2.25]
  7 days from the start of administration of this drug | 1.58 [1.11 to 2.25]
  14 days from the start of administration of this drug | 1.75 [1.24 to 2.45]
  21 days from the start of administration of this drug | 1.75 [1.24 to 2.45]
  28 days from the start of administration of this drug | 1.80 [1.29 to 2.52]

ADVERSE EVENTS:
Time Frame: From the start date of treatment with Paxlovid PACK to 28 days after the end of treatment, up to approximately 45days.
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | Paxlovid PACK (Nirmatrelvir/Ritonavir)
All-Cause Mortality (participants affected / at risk) | 16/2829
Serious Adverse Events (participants affected / at risk) | 51/2829
Other Adverse Events (participants affected / at risk) | 474/2829
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paxlovid PACK (Nirmatrelvir/Ritonavir) (N=2829)
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 2
Cholangitis acute (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia aspiration (Infections and infestations) | 10
Pneumonia bacterial (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Marasmus (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral venous thrombosis (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paxlovid PACK (Nirmatrelvir/Ritonavir) (N=2829)
Vertigo (Ear and labyrinth disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 92
Faeces soft (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 35
Oral discomfort (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 17
Malaise (General disorders) | 12
Oedema (General disorders) | 3
Pyrexia (General disorders) | 8
Hepatic function abnormal (Hepatobiliary disorders) | 5
Bronchitis (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 3
Pneumonia aspiration (Infections and infestations) | 4
Pneumonia bacterial (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 5
Blood pressure decreased (Investigations) | 5
Fibrin D dimer increased (Investigations) | 3
Liver function test increased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 18
Dehydration (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 5
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 189
Headache (Nervous system disorders) | 6
Olfactory dysfunction (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 4
Taste disorder (Nervous system disorders) | 48
Delirium (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 14
Rash pruritic (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT05263908/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT05263908/SAP_001.pdf